CLINICAL TRIAL: NCT00502957
Title: Biofeedback for Functional Constipation: Efficacy and Predictive Factors of Success
Brief Title: Biofeedback Treatment for Functional Constipation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H9654-26326
Record Dates: First submitted 2007-07-16; First posted 2007-07-18 (Estimated); Last update posted 2010-06-25 (Estimated); Status verified 2009-08

CONDITIONS: Constipation
Keywords: biofeedback; constipation
MeSH Terms: conditions — Constipation | interventions — Biofeedback, Psychology

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Biofeedback

SUMMARY:
The purpose of this randomized, controlled trial is to examine how well biofeedback treatment works to improve constipation. The study is comparing two kinds of biofeedback treatment: 1) anorectal-specific biofeedback therapy and 2) generalized biofeedback therapy using relaxation techniques.

The study will also examine which medical and psychological factors determine biofeedback success for treating constipation, such as bowel habits, emotional reactions to constipation, and levels of stress and psychological distress.

DETAILED DESCRIPTION:
This is a randomized controlled trial (RCT) to evaluate the efficacy of anorectal biofeedback therapy for functional constipation secondary to pelvic floor dyssynergia. Participants will be randomized to either six sessions of anorectal biofeedback or to six sessions of generalized biofeedback.

Participants will complete questionnaires at baseline, at completion of randomized treatment(12 weeks), and six months after completion of treatment to measure change in bowel habits, constipation severity, constipation-related quality of life, and constipation-related disability. An examination of psychosocial factors will also be conducted prior to treatment to distinguish which ones are predictive of biofeedback success for functional constipation.

ELIGIBILITY:
Inclusion Criteria:

* chronic constipation
* medical recommendation to undergo biofeedback training

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2005-03; Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Madhulika G Varma, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

REFERENCES:
- [Derived] Hart SL, Lee JW, Berian J, Patterson TR, Del Rosario A, Varma MG. A randomized controlled trial of anorectal biofeedback for constipation. Int J Colorectal Dis. 2012 Apr;27(4):459-66. doi: 10.1007/s00384-011-1355-9. Epub 2011 Dec 9. PMID 22159695